CLINICAL TRIAL: NCT04802239
Title: Assessment in Healthy Volunteers of the Analgesic Effect Monitored by the NOL Index of a Hypnotherapy Session Versus a Calm Waking State During Standardized Thermal Harmful Stimulation. The HYPTHENOL Study
Brief Title: Assessment in Healthy Volunteers of the Analgesic Effect Monitored by the NOL Index During Hypnotherapy Session
Acronym: HYPTHENOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, MD,Ph D ,Professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2021-2542
Record Dates: First submitted 2021-03-01; First posted 2021-03-17 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Pain; Hypnosis
Keywords: health volunteers; hypnosis; pain; NOL index; Bi spectral index
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective monocentric trial randomized to "cross-over". Each subject is its own witness, in the comparison of the analgesic effect of a hypnotherapy session versus a calm waking state, during standardized stimulation with monitoring of the NOL noxious index. As each of the subjects will be subjected to the two aforementioned states, a minimum time of 48 hours will be observed between the two exposures (hypnotherapy or calm watch) to reduce the memorization and the sensitization generated by the thermal stimulation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Prospective monocentric trial randomized to "cross-over". Each subject is its own witness, in the comparison of the analgesic effect of a hypnotherapy session versus a calm waking state, during standardized stimulation with monitoring of the NOL noxious index. As each of the subjects will be subjected to the two aforementioned states, a minimum time of 48 hours will be observed between the two exposures (hypnotherapy or calm watch) to reduce the memorization and the sensitization generated by the thermal stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calm waking group (Active Comparator): calm waking state group
  Interventions: Other: calm wake group
- hypnosis session (Experimental): hypnosis session group
  Interventions: Other: Medical hypnosis group

INTERVENTIONS:
Other: Medical hypnosis group — Hypnotic induction is performed according to a standard protocol and identical for all.
  A script will be written to give all the important steps. .Only the pleasant place and the characteristics of the analgesic glove will be different between the subjects .the procedure will follow the following protocol:
  * State of calm at rest of 3 minutes.
  * Hypnotic induction by catalepsy of the eyes guided by breathing.
  * The hypnosis session takes place in safety place , with glove protect by dissociation and confusion techniques.
  Arms: hypnosis session
Other: calm wake group — healthy volunteers will observe 3 minutes calm waking state before standardized thermal harmful stimulation
  Arms: calm waking group

SUMMARY:
to evaluate, in healthy volunteers, the analgesic effect of medical hypnosis versus a state of calm watch during a thermal harmful stimulation and monitored by a quantitative, objective criterion and validated in the literature that is the NOL index .Monitoring the NOL index will allow us to assess the level of nocipception linked to standardized thermal stimulation between the two states: hypnotherapy versus calm watch state. Each subject of the study will be subject to the two conditions (hypnosis versus calm watch state) during which participant will be subjected to the same type of thermal stimulation with the same monitoring of the parameters under study.

The choice, for each subject, to start with the hypnosis session versus the calm standby session will be decided by randomization according to the "cross-over" drawing of this study, and before session 1.

Using the NOL index, the investigators want to check what is the real and objective impact of hypnosis on the pain induced by a standardized harmful stimulus.

If the investigators find a significant difference in the variations of the NOL index after harmful stimulation between the two situations (hypnosis versus calm watch state) then the investigators can offer this monitoring in future studies, to follow the induced hypnotic trance in patients with local anesthesia during surgery associated with hypnosedation.

DETAILED DESCRIPTION:
Study desing: Monocentric, prospective randomized test in "crossover" (each subject being its own witness), comparing the analgesic effect of a hypnotherapy session versus a calm standby state.

Population studied: Healthy volunteers, adults Sample size: 12 subjects will be included in total, each one being subjected to the two sessions with different conditions (hypnosis versus calm watch state) subjects will be evaluated and classified by the hypnotisability score of the Harvard group scale of hypnotic susceptibility form A (HGSHS: A) translated into French by Hernan A and J Becchio

Participants will be classified into 4 groups :

i)Highly hypnotizable group (10-12), ii) Moderately hypnotizable group (7-9) iii)Slightly hypnotizable group (3-6) iv)Little hypnotizable group (0-2) The first two groups (score of 7 and more) will be included in the experimental study.Evaluation will be carried out according to 2 states over 2 different days, with a minimum interval between the two sessions of 48 hours.State of calm watch with thermal stimulation = control condition (session 1 or 2 depending on randomization).State of hypnotic trance with thermal stimulation and associated with hypnotic analgesic suggestions = experimental condition (session 1 or 2 depending on randomization).Thermal stimulation is performed using a Thermo Q-sense thermal probe (Medoc Advanced Medical Systems, Israel). The probe will first be calibrated before contact with the subject. Then, the probe will be placed on the palm side of the left hand for all subjects and during the two sessions (calm and hypnosis).This probe has already been used by our team for other research work and is completely safe, causing no skin damage to the subject. The Department of Anesthesiology and Pain Medicine owns this device. The temperature varies between 30 ° to 50 ° C in about 30 seconds, and stops under three conditions: when the subject clicks on a controller, at his requests, or when this temperature reaches 50 ° C.The NOL index: the NOL will be recorded continuously through the PMD200TM monitor, available at HMR in current clinical practice of anesthesia. Registration will begin at the start of sessions and procedures. PMD200TM also records heart rate values automatically.Sedline (EEG monitor peranesthesia, Masimo, CA, USA) will also be connected to the subject to assess the spectrogram of EEG waves (electroencephalography) with or without hypnosis. This monitor is non-invasive and gives its parameters using an electrode that sticks to the subject's forehead. These monitors are used in common clinical anesthesia practice and are available and used at HMR.The data will be electronically exported at the end of the experiment in a completely anonymous manner and kept in confidential, anonymous and protected electronic files of the study for a period of 7 years.

A pre-hypnosis consultation with the subjects will take place just before the session in order to harvest a place of safety and , assess its major communication channel, collect useful information for the realization of the "analgesic glove", establish a signal with him to rule on the state of trance and answer their questions.Even if the protocol is standard in its design, the protocol remains specific to each participant and adapted to the place of "safe place" and / or to the characteristics of the protective glove or "analgesic glove" that participant has chosen.

A formal hypnosis session will be conducted on the theme of a safety location chosen by the subject. When the trance is confirmed, the investigators will carry out the thermal stimulation starting at 30 ° C, and increasing the temperature until the stop requested by the subject (via a controller, or by its request). To stay safe, stimulation by this thermal probe cannot exceed 50 ° C over 30 seconds, and therefore cannot cause any burn. The technique of "antalgic suggestion" will be done through a protective glove and an analgesic cream, which will modulate the pain. Hypnotic induction is performed according to a standard protocol and identical for all. A script will be written to give all the important steps. This is a semi-structured hypnosis which will follow an identical pattern from one subject to another.Only the pleasant place and the characteristics of the analgesic glove will be different between the subjects because they are personal choices. This is important to keep a permissiveness in hypnosis and to adapt it to each subject according to the recommendations of permissive hypnosis.

the procedure will follow the following protocol:

* State of calm at rest of 3 minutes.- Hypnotic induction by catalepsy of the eyes guided by breathing.- The interview takes place in a place of safety, or leisure activity by dissociation and confusion techniques.- The place of security, this activity will be specific to each subject and will be personal.
* The analgesic suggestion will be made through a "protective glove".The hypnotic state will be considered to have been reached when the subject indicates it to the clinician using a previously installed signal and in response to three questions: "Are participants comfortable where they are ?"; "Did participants put the glove and the cream right on their hand ?";" Is the hand well protected ?".The hypnotic state is affirmed if the subject answers "yes" to the 3 questions. If the comfort of the subject is not satisfactory, the therapist will deepen the hypnotic trance with other suggestions, and will wait for the time necessary for the subject to reach this state. If, despite this, the subject cannot reach the desired state, the subject will be classified as resistant and will be analyzed as such.An objective evaluation of the trance signs will be made by an outside observer to note the presence or not of the following signs - immobility of the body- respiratory slowdown- slowdown in movements- slowing of responses and ideas: slowness of speech, and altered voice- variation in face color: pallor, redness- relaxed face muscles- modification of the overall muscle tone- gaze fixed- modified swallowing: slowed or accentuated- awakening behaviors at the end of the trance: blinking, rubbing of the eyes, yawning.An evaluation of the perception-pain score will be made with the subject at the end of the session: P0: no perception or pain, P1: perception but no pain, P2: perception and average pain, P3: perception and pain present, P4: severe pain perception

Regarding the "control" condition, i.e. without hypnosis :

* These are the same subjects of the study. - Participants will be put in a calm standby situation, at rest, in a dorsal decubitus, eyes closed for at least 3 minutes.
* The probe will deliver an increasing thermal intensity starting from 30 ° to a safe maximum of 50 ° in 30 seconds too.- An identical evaluation of the perception-pain score will be made with the participant at the end of the session.Statistical plan:According to previous studies carried out in our department, the variation of the NOL (delta-NOL) index following a harmful stimulation without analgesics is approximately 15 +/- 5. The use of an analgesic such as N2O made it possible to reduce this delta-NOL by approximately 35% (Richebé et al., in press in European Journal of Anaesthesia).

Believing that hypnotherapy could also reduce this delta-NOL by 40%, with an alpha to 0.05 and a power of 80% and a bilateral test, the number of subjects necessary to meet our main objective will be 12. The investigators do not expect a loss in follow-up during this study on healthy voluntary subjects. The investigators will therefore include a total of 12 participants who will have scanned> 6 on the aforementioned hypnotisability scale during screening.

Data analyzes :

Statistical analyzes will be carried out using version 9.4 or higher of SAS. The level of significance will be set at 0.05 bilaterally, unless otherwise indicated. Continuous data will be expressed on average or median with the appropriate dispersion index (standard deviation (SD) or interquartile range). The categorical data will be expressed in number with proportion. Confidence intervals (CI) will be expressed at a level of 95%. The normal distribution of continuous variables will be assessed using the Shapiro-Wilk test. The comparison of these variables will be carried out using Student's t test if the distribution is normal and using the Mann-Whitney non-parametric test otherwise. The categorical variables will be analyzed using the Khi-two test when the number of subjects in all groups is ≥ 5 and using the exact Fisher test otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ASA score I, II Age 18 or over

  * Acceptance of protocol and hypnosis in general
  * Good understanding of French
  * Agreement to comply with the recommendations of the protocol Score of the Stanford-Hildegard hypnotisability scale (HGSHS: A) >6

Exclusion Criteria:

* Psychiatric or neurological pathology making participation in the protocol difficult

  * Drug or alcohol consumption within 24 hours of the evaluation tests and the protocol
  * Analgic consumption within 24 hours before the test (tests and study)
  * Pregnant woman
  * Usual practice of sophrology, hypnosis, or meditation
  * Score of the Stanford-Hildegard hypnotisability scale (HGSHS: A) <6.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Delta Nol index ( no unit ) | From 1 minute before to 5 minutes after the Standard Thermal Stimulation (STS) for each subject
  Evaluate in healthy volunteers under hypnosis versus their own control in a calm state the variability of the NOL index (delta-NOL) which is the difference between the value of the peak (average of 3 values around the NOL peak) minus the basal pre-stimulation value, after standardized thermal stimulation

SECONDARY OUTCOMES:
Basal value of NOL index ( no unit ) | from 5 minutes to 1 minute before stimulation (STS)
  Evaluate in volunteers under hypnosis versus their own control (calm state) the basic level of the NOL
Peak value for NOL (no unit ) | from start to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) the peak value for NOL before and after stimulation STS
Area Under the Curve (AUC) for NOL (no unit) | from start to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) the AUC for NOL
Peak value of heart rate (HR ) (unit: beat per minute) | From 1 minute before to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) variation of HR before and after stimulation (STS)
Aera Under the Curve (AUC) of heart rate (HR ) (unit: beat per minute) | From 1 minute before to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) variation of HR before and after stimulation (STS)
Peak value of Mean Arterial Blood Pressure (MABP) (unit : mmHg) | From 1 minute before to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) variation of MABP before and after stimulation (STS)
Area Under the Curve (AUC) of Mean Arterial Blood Pressure (MABP) (unit : mmHg) | From 1 minute before to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) variation of MABP before and after stimulation (STS)
Peak value of Bispectral index ( BIS) ( no unit ) | from 1 minute to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) BIS index before and after stimulation (STS)
Area Under the Curve) of Bispectral index ( BIS) ( no unit ) | from 1 minute to 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) BIS index before and after stimulation (STS)
Pain scores (from 0 to 10 ) (no unit) | 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) the pain score
Pain perception (yes/no) | 5 minutes after stimulation (STS)
  Evaluate in healthy volunteers under hypnosis versus their own control (calm state) the pain perception
Hypnotic transe perception (yes/no) | 2 minutes before stimulation (STS)
  Assess only in the hypnosis group
Carry over effect (exposition order) (no unit) | from 1 minute before to 5 minutes after stimulation (STS)
  Evaluate variations in the NOL index according to the "carry-over effect" randomization range (order of exposure to hypnosis) during experimental stimulation (STS)
Peak value of NOL index (no unit) | from 1 minute before to 5 minutes after painful suggestion
  Evaluate variation of NOL index with painful suggestion in two state calm and hypnosis without stimulation STS
Area Under the Curve (AUC) of NOL index | from 1 minute before to 5 minutes after painful suggestion
  Evaluate variation of NOL index with painful suggestion in two state calm and hypnosis without stimulation STS

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de Montreal, Montreal, Quebec, Canada